CLINICAL TRIAL: NCT00684151
Title: Lipid-lowering Therapy in Patients With High Cardiovascular Risk and Their 3-year Mortality Rate in General Practice in Thailand
Brief Title: Survey of Lipid Goal Attainment and Mortality in Patients With High Cardiovascular Risk in Thailand
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CTH-DUM-2007/1
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Dyslipidemia
Keywords: Lipid-lowering
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with high cardiovascular risk who have been treated with lipid-lowering drugs at least 3 months

SUMMARY:
The first phase of the study is a hospital-based cross-sectional, epidemiological survey. The required sample size is 1,260 patients from 50 hospitals across Thailand. Each of the hospital will enroll 10 to 40 consecutive patients, depending on case availability on the date conducting the survey, with dyslipidemia and classified as high risk as defined by the protocol. Lipid levels will be based on serological analysis conducted by a local laboratory.

For the second phase, each subject will be followed for survival status at 36 months after enrollment. Such follow-up will be done by searching the Thai National Vital Event Registration Database using subjects' Population Identification Number. All activities regarding case selection and data collection will be done by well trained clinical research associates (CRAs). The CRAs are from Khon Kaen University where the Statistical Coordinating Center (SCC) for this project is based and are independent of the investigator. Random auditing visits will also be performed by auditors independent of the SCC. These are to ensure not only high quality data but also protecting right and well being of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of high cardiovascular risk
* Dyslipidemic currently being treated with the same therapy for at least 3 months

Exclusion Criteria:

* Recent major trauma(within 12 weeks)
* Recent surgery requiring anesthesia including coronary bypass graft(within 12 weeks)
* Acute or abrupt change(within 1 month) in usual diet
* Pregnancy, breast-feeding currently, or postpartum within the last 6 months

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high cardiovascular risk who have been treated with lipid-lowering drugs at least 3 months
Sampling Method: Non-Probability Sample
Enrollment: 1240 (Actual)
Dates: Start 2008-04; Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
LDL-cholesterol | June2008

SECONDARY OUTCOMES:
Survival | June 2011

CONTACTS AND LOCATIONS:
Overall Officials: Bandit Thinkhamrop, Ph.D, Study Director — Khon Kaen University; Songkwan Silaruks, M.D., Principal Investigator — Khon Kaen University
Locations (49):
- Thailand (49):
  - Research Site, Kannayao, Bangkok
  - Research Site, Maung, Changwat Ang Thong
  - Research Site, Maung, Changwat Chachoengsao
  - Research Site, Maung, Changwat Chai Nat
  - Research Site, Maung, Changwat Chanthaburi
  - Research Site, Maung, Changwat Chumphon
  - Research Site, Muang, Changwat Khon Kaen
  - Research Site, Maung, Changwat Krabi
  - Research Site, Maung, Changwat Lampang
  - Research Site, Maung, Changwat Lamphun
  - Research Site, Maung, Changwat Lop Buri
  - Research Site, Maung, Changwat Nan
  - Research Site, Muang, Changwat Nong Khai
  - Research Site, Maung, Changwat Nonthaburi
  - Research Site, Maung, Changwat Phangnga
  - Research Site, Maung, Changwat Phatthalung
  - Research Site, Maung, Changwat Phayao
  - Research Site, Maung, Changwat Phichit
  - Research Site, Maung, Changwat Phitsanulok
  - Research Site, Maung, Changwat Phrae
  - Research Site, Maung, Changwat Prachuap Khiri Khan
  - Research Site, Ban Pong, Changwat Ratchaburi
  - Research Site, Maung, Changwat Ratchaburi
  - Research Site, Maung, Changwat Rayong
  - Research Site, Maung, Changwat Roi Et
  - Research Site, Maung, Changwat Samut Sakhon
  - Research Site, Maung, Changwat Samut Songkhram
  - Research Site, Maung, Changwat Satun
  - Research Site, Maung, Changwat Si Sa Ket
  - Research Site, Hat Yai, Changwat Songkhla
  - Research Site, Maung, Changwat Suphan Buri
  - Research Site, Maung, Changwat Surat Thani
  - Research Site, Maung, Changwat Surin
  - Research Site, Maung, Changwat Tak
  - Research Site, Maung, Changwat Trang
  - Research Site, Maung, Changwat Ubon Ratchathani
  - Research Site, Maung, Changwat Udon Thani
  - Research Site, Maung, Chiang Mai
  - Research Site, Maung, Kamphaeng Phet H
  - Research Site, Maung, Kanchanaburi
  - Research Site, Maung, Mahasarakarm
  - Research Site, Muang, Nakhorn Phanom
  - Research Site, Maung, Nakorn Nayok
  - Research Site, Maung, Nokhon Si Thammarat
  - Research Site, Maung, Nokorn Pathom
  - Research Site, Maung, Phra Nakhon Si Ayutthaya
  - Research Site, Maung, Phuket
  - Research Site, Maung, Uthaithani
  - Research Site, Maung, Uttaradit